CLINICAL TRIAL: NCT07188220
Title: Perspectives on the Multidisciplinary Approach to Metabolic Dysfunction-associated Steatohepatitis: a Qualitative Study With Patients From the MASH-Cardiovascular Programme at Hospital de Sant Pau i la Santa Creu, Barcelona
Brief Title: Patients' Perspectives on Metabolic Dysfunction-associated Steatohepatitis: a Qualitative Study
Status: Recruiting | Type: Observational
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: 25/093 (OBS)
Record Dates: First submitted 2025-07-30; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-07

CONDITIONS: Metabolic Dysfunction Associated Steatohepatitis (MASH)
Keywords: Qualitative; MASH; MASLD; Perceptions; Semi-structured interviews

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this qualitative study is to explore and identify the expectations, perceptions, attitudes, needs, and knowledge related to the management of metabolic dysfunction-associated steatohepatitis (MASH) in patients diagnosed with this condition, before and after their participation in the MASH-Cardiovascular Programme at Hospital de la Santa Creu i Sant Pau, Barcelona.

The main research question is:

What expectations, attitudes, needs, and perceptions do patients with MASH participating in the MASH-Cardiovascular Programme exhibit before and after the intervention?

Participants will undergo two semi-structured interviews: one prior to, and one following, their involvement in the MASH-Cardiovascular Programme at Hospital de Sant Pau i la Santa Creu, Barcelona.

ELIGIBILITY:
Inclusion Criteria:

* Patients who voluntarily agree to participate in the MASH-Cardiovascular Programme.
* Patients followed in the outpatient hepatology/gastroenterology clinic at Hospital de Sant Pau with a diagnosis of MASH and fibrosis stage F2-F4.
* Patients aged between 18 and 75 years.
* Patients with a BMI ≥ 27 kg/m².
* Patients who consent to participate in the study-specific interviews.

Exclusion Criteria:

* Patients who do not agree to participate in the study-specific interviews.
* Patients meeting exclusion criteria of the MASH-Cardiovascular Programme:
* Patients with decompensated liver cirrhosis.
* Patients who are vegetarians or have dietary habits/preferences that prevent adherence to standard-of-care nutritional guidelines.
* Patients with moderate-to-severe alcohol consumption (>20 g/day for women and >40 g/day for men).
* Patients with an eGFR < 30 mL/min.
* Patients with malnutrition.
* Patients with type 1 diabetes or other forms of diabetes.
* Patients who are candidates for bariatric surgery.
* Patients with active malignancy.
* Patients with advanced or unstable heart failure.
* Patients with eating disorders or severe psychiatric illness.
* Patients currently enrolled in another clinical trial.
* Pregnant women or women planning to become pregnant.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Gender Based: Yes — The semi-structured interview includes a specific gender identity question: Which gender do you identify with?
  * Woman
  * Man
  * Non-binary
  * Prefer not to answer
Study Population: The study population will consist of individuals diagnosed with MASH who are referred to the multidisciplinary MASH-Cardiovascular Programme at Hospital de la Santa Creu i Sant Pau in Barcelona.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2025-06-03 (Actual); Primary Completion 2027-12-20 (Estimated); Study Completion 2028-01-20 (Estimated)

PRIMARY OUTCOMES:
Perceptions | At baseline (within two weeks before starting the programme) and at one-year follow-up (within two weeks before and after completing the programme)
  Perceptions explored through semi-structured interviews
Attitudes and expectatives | At baseline (within two weeks before starting the programme) and at one-year follow-up (within two weeks before and after completing the programme)
  Attitudes and expectatives explored through semi-structured interviews
MASH-related knowledge | At baseline (within two weeks before starting the programme) and at one-year follow-up (within two weeks before and after completing the programme)
  MASH-related knowledge explored through semi-structured interviews
Unmet needs | At baseline (within two weeks before starting the programme) and at one-year follow-up (within two weeks before and after completing the programme)
  Unmet needs explored through semi-structured interviews

CONTACTS AND LOCATIONS:
Locations (1):
- IR Sant Pau, Barcelona, Spain